CLINICAL TRIAL: NCT03921593
Title: Prospective Longitudinal Observational Study on Insulin Dependent Diabetic Patients Undergoing Any Form of Solid Organ Pancreas Transplantation Aimed to Clarify Quality of Life Changes After Pancreas Transplantation
Brief Title: Quality of Life in Pancreas Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 18/SC/0385
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus; Quality of Life
Keywords: quality of life; pancreas transplant
MeSH Terms: conditions — Diabetes Mellitus | interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Simultaneous Pancreas Kidney Transplant Recipients: Patient affected by Insulin Dependent Diabetes Mellitus and renal failure undergoing Simultaneous Pancreas Kidney Transplant (SPK)
  Interventions: Procedure: Solid Organ Pancreas Transplantation with or without Kidney Transplantation
- Pancreas after kidney Transplant Recipients: Patient affected by Insulin Dependent Diabetes Mellitus and renal failure undergoing Pancreas after kidney Transplant (PAK)
  Interventions: Procedure: Solid Organ Pancreas Transplantation with or without Kidney Transplantation
- Pancreas Transplant Alone Recipients: Patient affected by Insulin Dependent Diabetes Mellitus with hypoglycemia unawareness undergoing Pancreas Transplant Alone (PTA)
  Interventions: Procedure: Solid Organ Pancreas Transplantation with or without Kidney Transplantation

INTERVENTIONS:
Procedure: Solid Organ Pancreas Transplantation with or without Kidney Transplantation — Deceased donor pancreas transplantation

SUMMARY:
Quality of Life for individuals with Insulin Dependent Diabetes Mellitus (IDDM) can be severely impaired by acute and chronic complications of the disease.

Solid organ pancreatic transplantation restores endocrine pancreatic function. However, it is also burdened by high perioperative morbidity and mortality.

Clinical benefits and risks of this intervention have been extensively clarified, but our knowledge about quality of life gain, often mentioned among the assets of transplantation, is still limited.

This study aims to quantify the impact of all forms of Solid Organ Pancreas Transplantation on quality of life (QOL).

DETAILED DESCRIPTION:
Rationale of the study:

There are 3.5 million people in the United Kingdom diagnosed with diabetes. Their life expectancy is significantly reduced when compared to non-diabetic population. The long standing poor metabolic control causes a cluster of complications such as metabolic instability, cardiovascular disease, nephropathy, retinopathy and neuropathy which have a major impact on the clinical and social wellbeing of these individuals.

Solid organ pancreatic transplantation restores endocrine pancreatic function, but it is still burdened by significant perioperative morbidity and mortality.

There are other less invasive transplant options we can offer to this cohort of patients. The most common are Kidney Transplant Alone (KTA) from deceased or living donor in the diabetic and uremic patients and Islets Transplant (IT) for those with hypoglycemia unawareness and preserved renal function.

Although current literature suggests that the less invasive approaches may be less effective in the long term, potentially they could resolve the most compelling clinical needs at a lower surgical risk.

There is now a general consensus that the surgical risks of pancreatic solid organ transplantation must be weighed against clinical outcomes as well as QOL gain

Aims of the study:

This study aims to quantify QOL trajectory pre- and post- pancreas transplantation and identify correlations between QOL and clinical outcomes. The data collected will be utilized to understand which forms of solid organ pancreas transplantation are associated with greater/ lesser QOL gain and to compute a cost effectiveness analysis of this intervention.

Methods:

The core of the study will be a prospective quasi-experimental design focusing on QOL outcomes for patients on the pancreas transplant waiting-list at Oxford University Transplant Centre.

Patients active on the Oxford Transplant Centre Pancreas Transplant Waiting list will be invited to take part to this study.

Participants will be requested to complete one set of validated generic and disease specific (diabetes and kidney failure where applicable) QOL questionnaires pre-transplantation and at three time points post-transplantation: 6 weeks, 6 months and 1 year. The research team will collect clinical and hospital usage data at the same time points.

At the end of data collection, statistical analysis will aim to discern overall QOL changes in terms of Quality Adjusted Life Years (QALY), but also whether different cohorts of pancreas transplant recipients (SPK, PAK, and PTA) have different QOL outcomes and in which domains of QOL they differ.

A cohort of patients who receive a PT will be matched to a cohort of patients who remain on the PT waiting-list. Matching estimators, including Propensity Score and Coarsened Exact Matching, will be used to achieve covariate balance between the synthetic treated and control groups in order to estimate the causal effect of QoL changes post-transplantation.

Cumulative hospital costs of care by treatment group will be analysed using appropriate regression methods for non-normal, continuous outcomes. Continuous QOL outcomes will be analysed using generalised linear models.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Insulin Dependent Diabetic Patients
* Active on Pancreas Transplant Wait List

Exclusion Criteria:

* Not fluent in English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Insulin Dependent diabetic adult patients with either renal failure or hypoglycemia unawareness or both, active on Oxford transplant centre pancreas transplant waiting list and fluent in English
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2018-11-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of Quality of Life | pre-transplantation, 6/52 post transplantation, 6/12 post transplantation, 1 year post transplantation
  Completion of EQ-5D-5L questionnaire. Scoring rules Each Dimension has 5 possible levels: 1 no problems, 2 slight problems, 3 moderate problems, 4 severe problems, 5 and extreme problems.
  Each level corresponds to a 1-digit code: 1-2-3-4-5. The final score is a 5-digit code describing the responder health state. These numbers have no arithmetic properties and should not be used as cardinal scores.
  Each 5-digit combination correspond to a possible health state. A total of 3125 possible health states is defined in this way. For example, state 11111 indicates no problems on any of the 5 dimensions, while state 12345 indicates no problems with mobility, slight problems with washing or dressing, moderate problems with doing usual activities, severe pain or discomfort and extreme anxiety or depression.
Quantification of Quality of Life | pre-transplantation, 6/52 post transplantation, 6/12 post transplantation, 1 year post transplantation
  Completion of Diabetes Quality of Life questionnaire (DQOL) DQOL includes 46 core items forming four scales targeted at particular health-related concerns of individuals with Insulin Dependent Diabetes Mellitus, a generic health item that does not contribute to the scales Scoring rules Dimensions and DQoL total scores (average score across the 4 dimensions) are scored 0-100, where 0 is the lowest possible quality of life and 100 the highest.
Quantification of Quality of Life | pre-transplantation, 6/52 post transplantation, 6/12 post transplantation, 1 year post transplantation
  Completion of Kidney Disease Quality of Life Short Form questionnaire (KDQOL-SF) KDQOL-SFTM includes multi-item scales targeted at particular health-related concerns of individuals with kidney disease and generic scales derived from the short form 36 (SF-36),Scoring Rules
  1) Each possible response for each item corresponds to a pre-coded numeric value. 2) The raw pre-coded numeric values are transformed to a 0-100 range, with higher transformed scores reflecting better quality of life ( the lowest and highest possible scores are 0 and 100, respectively ).
  3) Items on the same scale are averaged to ether to create the scale scores. Items that are left blank are not take into account: the final score for each scale represents the average for all the items in that scale that the respondent answered.
Quantification of Quality of Life | pre-transplantation, 6/52 post transplantation, 6/12 post transplantation, 1 year post transplantation
  Completion of Short Form 12 v.2 questionnaire (SF-12 v.2®) includes 8 domains and 12 items that form two Components: Physical Health Component (PCS) and Mental Health Component (MCS) A computer-based scoring algorithm is used to calculate scores: Physical Component Summary (PCS) and Mental (MCS) Component Summary scales are generated using norm-based methods. Scores are transformed to have a mean value of 50, standard deviation (SD) 10, where scores above or below 50 are above or below average physical or mental well-being, respectively.

SECONDARY OUTCOMES:
Correlation between clinical status and quality of life pre-transplantation | pre-transplantation, 6/52 post transplantation, 6/12 post transplantation, 1 year post transplantation
  Identification of which clinical phenotypes correspond to higher quality of life scores collection of clinical data at the same time points as quality of life questionnaires to establish correlation/causal effect between clinical and qol data
Estimate cost-effectiveness of pancreas transplantation | pre- transplant, 1 year
  calculation of Quality Adjusted Life Years (QALYs) As per NICE recommendation, utility scores derived by EQ5D5L will be used to calculate Quality Adjusted Life Years before transplantation and at one year from transplant to calculate QALY gain after pancreas transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Friend, MA, MB, FRCS, MD, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospital NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Quality and Outcomes Framework (2014/15), Diabetes Prevalence Model 2016 (Public Health England) and 2012 APHO Diabetes Prevalence Model.
- [Background] 2. Livingstone, S.J. et al (2015) Estimated Life Expectancy in a Scottish Cohort with Type 1 Diabetes, 2008-2010. JAMA 313(1) 37-44 78 Seshasai SR on behalf of the Emerging Risk Factors Collaboration (2011) Diabetes mellitus, fasting glucose, and risk of cause-specific death. N Engl J Med. 3;364(9):829-41
- [Background] Diabetes mellitus: a major risk factor for cardiovascular disease. A joint editorial statement by the American Diabetes Association; The National Heart, Lung, and Blood Institute; The Juvenile Diabetes Foundation International; The National Institute of Diabetes and Digestive and Kidney Diseases; and The American Heart Association. Circulation. 1999 Sep 7;100(10):1132-3. doi: 10.1161/01.cir.100.10.1132. No abstract available. PMID 10477541
- [Background] Liew G, Michaelides M, Bunce C. A comparison of the causes of blindness certifications in England and Wales in working age adults (16-64 years), 1999-2000 with 2009-2010. BMJ Open. 2014 Feb 12;4(2):e004015. doi: 10.1136/bmjopen-2013-004015. PMID 24525390
- [Background] Dean PG, Kukla A, Stegall MD, Kudva YC. Pancreas transplantation. BMJ. 2017 Apr 3;357:j1321. doi: 10.1136/bmj.j1321. PMID 28373161
- [Background] Taber DJ, Meadows HB, Pilch NA, Chavin KD, Baliga PK, Egede LE. Pre-existing diabetes significantly increases the risk of graft failure and mortality following renal transplantation. Clin Transplant. 2013 Mar-Apr;27(2):274-82. doi: 10.1111/ctr.12080. Epub 2013 Feb 6. PMID 23383719
- [Background] Lablanche S, Borot S, Wojtusciszyn A, Bayle F, Tetaz R, Badet L, Thivolet C, Morelon E, Frimat L, Penfornis A, Kessler L, Brault C, Colin C, Tauveron I, Bosco D, Berney T, Benhamou PY; GRAGIL Network. Five-Year Metabolic, Functional, and Safety Results of Patients With Type 1 Diabetes Transplanted With Allogenic Islets Within the Swiss-French GRAGIL Network. Diabetes Care. 2015 Sep;38(9):1714-22. doi: 10.2337/dc15-0094. Epub 2015 Jun 11. PMID 26068866
- [Background] White SA, Shaw JA, Sutherland DE. Pancreas transplantation. Lancet. 2009 May 23;373(9677):1808-17. doi: 10.1016/S0140-6736(09)60609-7. PMID 19465236